CLINICAL TRIAL: NCT02589470
Title: COMET Study Effectiveness of a Cognitive Remediation Program of Memory in Patients With Temporal Lobe Epilepsy
Brief Title: COMETE Study : COgnitive Rehabilitation of MEmory in Temporal Epilepsy
Acronym: COMETE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: CHU de Reims (Other); University Hospital, Strasbourg, France (Other); Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-a00733-46
Record Dates: First submitted 2015-10-16; First posted 2015-10-28 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Epilepsy
Keywords: cognitive rehabilitation; memory; epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COMETE (Experimental): patients will attend a specific rehabilitation programme of memory
  Interventions: Other: COMETE
- CONTROL (No Intervention): the control group where patients will benefit from a standard treatment

INTERVENTIONS:
Other: COMETE — Patients of COMETE group will attend 12 individual sessions of cognitive rehabilitation, which are not systematic in usual treatment, and will receive memory exercises via internet to continue cognitive exercizes at home.
  Arms: COMETE

SUMMARY:
Studies on the cognitive function have highlighted promising results concerning attention. In contrast, in the field of memory, the single cohort study that has been carried out, has not been randomised, with non comparable groups, the significant outcomes are therefore to be balanced.

In this study, patients with focal and structural temporal lobe epilepsy will be randomised in 2 groups : the COMETE group where patients will attend a specific rehabilitation programme of memory and the control group where patients will benefit from a standard treatment.

DETAILED DESCRIPTION:
Epilepsy is a chronic neurological disease among the most frequent ones. It causes cognitive disorders in 20 to 50 percent of patients with structural epilepsy, that is to say in connexion with an identified or presumed cerebral lesion. Compared to seizures, these cognitive disorders are a major additional factor of professional, social or family disability. They are particularly prevalent (50%) in temporal lobe epilepsy and preferentially affect language memory and abilities. These disorders are well described, they are multifactorial but no (drug and/or non drug) therapy has been validated yet.

Recently, techniques of cognitive rehabilitation have shown benefits in some neurological diseases, like multiple sclerosis.

Concerning adulthood epilepsy, the few cognitive rehabilitation studies that have been conducted present huge methodological gaps limiting the scope of theirs results.

Studies on the cognitive function have highlighted promising results concerning attention. In contrast, in the field of memory, the single cohort study that has been carried out, has not been randomised, with non comparable groups, the significant outcomes are therefore to be balanced.

Thus, in this study, patients with focal and structural temporal lobe epilepsy will be randomised in 2 groups : the COMETE group where patients will attend a specific rehabilitation programme of memory and the control group where patients will benefit from a standard treatment.

Work's hypothesis would be that patients undergoing the rehabilitation programme would present improved learning abilities (with impact on their memory performances) compared to patients with standard treatment.

This hypothesis is based on underlying theories of cognitive rehabilitation. This method predicts that by reinforcing some cognitive abilities that transfer to others, the improved learning abilities will also result in improved abilities in immediate memory, work memory, but will have no effect on verbal inhibition abilities, which will constitute a specific marker/indicator ? for the intervention. Moreover, patient care may have an impact on their quality of life and mood which are predictive factors for a good social and professional integration: that's why these indexes/criteria have to be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adults with structural temporal lobe epilepsy, according to Fischer et al (2005) criteria.
* Patients aged 18-70
* Patients with epilepsy for more than 2 year
* Patients with mild to severe memory impairment (minimum score : -1,6σ / average at Buschke Reminding Test, learning index
* Patients with equal or higher Intellectual Quotient than 70 (WAIS-IV)
* stabilized anti epileptic treatment (same treatment for the last 6 months)
* Patient who has given informed consent in writing
* Patients with social insurance
* Patients with internet connexion for weekly training at home

Exclusion Criteria:

* other progressive associated neurological (history of stroke for example) or psychiatric disease
* temporal lobe surgery within following 12 months
* presence of a progressive brain lesion
* legally protected adults or adults incapable of giving informed consent
* persons who are deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03-03 (Actual); Primary Completion 2019-09-03 (Estimated); Study Completion 2021-01-03 (Estimated)

PRIMARY OUTCOMES:
Buschke Reminding Test, learning index | 20 minutes
  this is a task of verbal memory : neuropsychologist read a list of 15 words, and patient must repeat a maximum of them

SECONDARY OUTCOMES:
digit span | 5 minutes
  this is a task of immediate memory : neuropsychologist read digit, and subject must recall them in the same order
Visual memory task | 10 minutes
  this is a task of visual memory : subject must memorize a grid
verbal fluencies | 5 minutes
  The performance measure is the total number of words that patient give in two minutes. there is two conditions : phonological condition : patient must recall words that start with the letter P; semantic condition : patient must recall words from animal category
Attentional tasks (TEA Battery) | 10 minutes
  This is attentional task on computer
Beck Depression Inventory | 10 minutes
  this is an inventory of depression

CONTACTS AND LOCATIONS:
Overall Officials: jean pierre VIGNAL, DR, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Service de Neurologie, Hôpital Central, CHRU de Nancy, Nancy, Lorraine, France

REFERENCES:
- [Background] Brissart H, Daniel F, Morele E, Leroy M, Debouverie M, Defer GL. [Cognitive rehabilitation in multiple sclerosis: a review of the literature]. Rev Neurol (Paris). 2011 Apr;167(4):280-90. doi: 10.1016/j.neurol.2010.07.039. Epub 2010 Dec 21. French. PMID 21176930
- [Result] Brissart H, Leroy M, Morele E, Baumann C, Spitz E, Debouverie M. Cognitive rehabilitation in multiple sclerosis. Neurocase. 2013;19(6):553-65. doi: 10.1080/13554794.2012.701644. Epub 2012 Aug 1. PMID 22853712